CLINICAL TRIAL: NCT00943306
Title: A Phase III, Long Term, Open Label, Follow on Study of Microsomal Triglyceride Transfer Protein (MTP) Inhibitor 'Lomitapide' (LOMITAPIDE) in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Long Term, Follow-on Study of Lomitapide in Patients With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEGR-733-012
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Familial Hypercholesterolemia
Keywords: Homozygous; Familial; Hypercholesterolemia; MTP; Apheresis; lomitapide; Homozygous Familial Hypercholesterolemia (HoFH)
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lomitapide (Experimental): Maximum tolerated dose of lomitapide in addition to existing lipid lowering therapy including plasmapheresis or lipid apheresis.
  Interventions: Drug: lomitapide

INTERVENTIONS:
Drug: lomitapide — 5-60 mg po every day
  Other Names: AEGR-733; BMS-201038

SUMMARY:
This was a long term follow on study to assess the continued long term safety and efficacy of lomitapide in patients with homozygous familial hypercholesterolemia.

DETAILED DESCRIPTION:
This was a phase III open label clinical trial to evaluate the long-term efficacy and safety of lomitapide at the maximum tolerated dose (for each patient) established during the clinical trial 733-005/UP1002. Subjects completing the 78-week treatment period in study 733-005/UP1002 who have not met any of the stopping criteria will be eligible to participate in 733-012. The treatment period continued until a decision was made by the local competent authority regarding marketing authorization. Lomitapide will be given orally once daily. Patient specific doses will be carried forward from 733-005/UP1002, but will not exceed the maximum tolerated dose the patient received during 733-005 /UP1002. The maximum dose for any patient was 80 mg/day. There was no reference therapy in this trial. The effects of the study drug were compared to baseline data (from 733-005/UP1002). Concomitant lipid-lowering therapy including plasmapheresis or LDL apheresis is permitted.

Note that hereafter, Week 0 in Study 733-005/UP1002 will be referred to as Baseline and Week 48 in Study AEGR-733-012 will be referred to as Week 126 (of overall treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Completed UP1002 or 733-005.
2. Willing and able to provide consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Met any of the stopping rules for study discontinuation at the final visit of study UP1002 or 733-005.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2012-09-17 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania; Mark Sumeray, MD, Study Chair — Aegerion Pharmaceuticals, Inc.
Locations (10):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - Robarts Research Institute, London, Ontario
  - Lipid Clinic and University of Montreal Community Genomic Medicine Center, Chicoutimi, Quebec
- Italy (4):
  - Medicina Interna Universitaria, Ferrara, Sicily
  - Dipartimento di Medicina Clinica e Delle Patologie Emergenti, Palermo, Sicily
  - Centro Universitario Dislipidemie, Milan
  - DAI Ematologia, Oncologia, Anatomia Patologica e Medicina, Roma
- South Africa (2):
  - Cardiology Research, Bloemfontein
  - University of Capetown, Cape Town

REFERENCES:
- [Background] Cuchel M, Bloedon LT, Szapary PO, Kolansky DM, Wolfe ML, Sarkis A, Millar JS, Ikewaki K, Siegelman ES, Gregg RE, Rader DJ. Inhibition of microsomal triglyceride transfer protein in familial hypercholesterolemia. N Engl J Med. 2007 Jan 11;356(2):148-56. doi: 10.1056/NEJMoa061189. PMID 17215532
- [Background] Cuchel M, Meagher E, Marais AD, et.al. Abstract 1077: A phase III study of microsomal triglyceride transfer protein inhibitor lomitapide (AEGR-733) in patients with homozygous familial hypercholesterolemia: interim results at 6 months. Circulation, Nov 2009; 120: S441
- [Derived] Larrey D, D'Erasmo L, O'Brien S, Arca M; Italian Working Group on Lomitapide. Long-term hepatic safety of lomitapide in homozygous familial hypercholesterolaemia. Liver Int. 2023 Feb;43(2):413-423. doi: 10.1111/liv.15497. Epub 2022 Dec 30. PMID 36520008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lomitapide
Started | 19
Completed | 16
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Sponsor decision due to non-compliance | 1

BASELINE CHARACTERISTICS:
Population: Baseline from initiation of treatment in Study 733-005/UP1002 (Safety Population)
Arm/Group | Lomitapide
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 2
  United States | 3
  South Africa | 9
  Italy | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -45.5 (31.35)

2. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent change in Low Density Lipoprotein Cholesterol (LDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: Safety Population - The number of patients in the Safety Population at time points after Week 126 decreased because the study remained active within each country until either approval of the marketing application was obtained, or, in countries where marketing authorization was not sought for, patients transitioned into an Expanded Access Program.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -51.0 (16.03)

3. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent change in Low Density Lipoprotein Cholesterol (LDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -58.5 (24.25)

4. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent change in Low Density Lipoprotein Cholesterol (LDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -60.1 (18.51)

5. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent change in Low Density Lipoprotein Cholesterol (LDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -74.0 (19.10)

6. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Percent change in Low Density Lipoprotein Cholesterol (LDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -51.1 (10.11)

7. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change in Total Cholesterol from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -43.2 (25.35)

8. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change in Total Cholesterol from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -46.9 (15.21)

9. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change in Total Cholesterol from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -51.0 (21.34)

10. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change in Total Cholesterol from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -54.1 (16.88)

11. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change in Total Cholesterol from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -65.2 (15.97)

12. Secondary Outcome: Percent Change in Total Cholesterol
Description: Percent change in Total Cholesterol from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -43.9 (5.01)

13. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B)
Description: Percent change in Apolipoprotein B (Apo B) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -53.6 (23.74)

14. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B)
Description: Percent change in Apolipoprotein B (Apo B) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -59.4 (12.60)

15. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B)
Description: Percent change in Apolipoprotein B (Apo B) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -65.1 (20.72)

16. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B)
Description: Percent change in Apolipoprotein B (Apo B) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -65.9 (15.76)

17. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B)
Description: Percent change in Apolipoprotein B (Apo B) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -76.7 (16.09)

18. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B)
Description: Percent change in Apolipoprotein B (Apo B) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -60.9 (12.17)

19. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change in Triglycerides from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -37.5 (42.52)

20. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change in Triglycerides from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -31.7 (37.09)

21. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change in Triglycerides from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -27.6 (48.88)

22. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change in Triglycerides from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -41.9 (33.16)

23. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change in Triglycerides from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -48.5 (34.24)

24. Secondary Outcome: Percent Change in Triglycerides
Description: Percent change in Triglycerides from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | 29.2 (58.74)

25. Secondary Outcome: Percent Change in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent change in Non High Density Lipoprotein Cholesterol (Non-HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -47.1 (27.83)

26. Secondary Outcome: Percent Change in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent change in Non High Density Lipoprotein Cholesterol (Non-HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -53.5 (16.42)

27. Secondary Outcome: Percent Change in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent change in Non High Density Lipoprotein Cholesterol (Non-HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -57.0 (24.07)

28. Secondary Outcome: Percent Change in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent change in Non High Density Lipoprotein Cholesterol (Non-HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -58.8 (17.73)

29. Secondary Outcome: Percent Change in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent change in Non High Density Lipoprotein Cholesterol (Non-HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -71.5 (17.65)

30. Secondary Outcome: Percent Change in Non High Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent change in Non High Density Lipoprotein Cholesterol (Non-HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -46.6 (5.19)

31. Secondary Outcome: Percent Change in Very Low Density Lipoprotein Cholesterol (VLDL-C)
Description: Percent change in Very Low Density Lipoprotein Cholesterol (VLDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -36.8 (43.90)

32. Secondary Outcome: Percent Change in Very Low Density Lipoprotein Cholesterol (VLDL-C)
Description: Percent change in Very Low Density Lipoprotein Cholesterol (VLDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -31.5 (36.32)

33. Secondary Outcome: Percent Change in Very Low Density Lipoprotein Cholesterol (VLDL-C)
Description: Percent change in Very Low Density Lipoprotein Cholesterol (VLDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -26.3 (49.94)

34. Secondary Outcome: Percent Change in Very Low Density Lipoprotein Cholesterol (VLDL-C)
Description: Percent change in Very Low Density Lipoprotein Cholesterol (VLDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -41.4 (34.20)

35. Secondary Outcome: Percent Change in Very Low Density Lipoprotein Cholesterol (VLDL-C)
Description: Percent change in Very Low Density Lipoprotein Cholesterol (VLDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -48.7 (33.41)

36. Secondary Outcome: Percent Change in Very Low Density Lipoprotein Cholesterol (VLDL-C)
Description: Percent change in Very Low Density Lipoprotein Cholesterol (VLDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | 30.6 (59.94)

37. Secondary Outcome: Percent Change in Lp(a)
Description: Percent change in Lp(a) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | 5.5 (43.62)

38. Secondary Outcome: Percent Change in Lp(a)
Description: Percent change in Lp(a) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | 10.2 (60.64)

39. Secondary Outcome: Percent Change in Lp(a)
Description: Percent change in Lp(a) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -12.8 (49.00)

40. Secondary Outcome: Percent Change in Lp(a)
Description: Percent change in Lp(a) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 13
Percent Change | 3.4 (54.22)

41. Secondary Outcome: Percent Change in Lp(a)
Description: Percent change in Lp(a) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -6.6 (48.99)

42. Secondary Outcome: Percent Change in Lp(a)
Description: Percent change in Lp(a) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -10.4 (35.64)

43. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change in High Density Lipoprotein Cholesterol (HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -8.3 (19.28)

44. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change in High Density Lipoprotein Cholesterol (HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | 3.8 (26.51)

45. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change in High Density Lipoprotein Cholesterol (HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -2.7 (21.22)

46. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change in High Density Lipoprotein Cholesterol (HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -12.5 (19.17)

47. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change in High Density Lipoprotein Cholesterol (HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -10.3 (27.68)

48. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change in High Density Lipoprotein Cholesterol (HDL-C) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -23.5 (2.27)

49. Secondary Outcome: Percent Change in Apolipoprotein AI (Apo AI)
Description: Percent change in Apolipoprotein AI (Apo AI) from Baseline (Week 0 of Study 733-005/UP1002) to Week 126 (Week 48 in Study AEGR-733-012).
Time Frame: Baseline and Week 126
Population: Week 126 Completers Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 17
Percent Change | -14.0 (17.71)

50. Secondary Outcome: Percent Change in Apolipoprotein AI (Apo AI)
Description: Percent change in Apolipoprotein AI (Apo AI) from Baseline (Week 0 of Study 733-005/UP1002) to Week 174 (Week 96 in Study AEGR-733-012).
Time Frame: Baseline and Week 174
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 16
Percent Change | -8.2 (20.12)

51. Secondary Outcome: Percent Change in Apolipoprotein AI (Apo AI)
Description: Percent change in Apolipoprotein AI (Apo AI) from Baseline (Week 0 of Study 733-005/UP1002) to Week 222 (Week 144 in Study AEGR-733-012).
Time Frame: Baseline and Week 222
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Percent Change | -2.7 (33.30)

52. Secondary Outcome: Percent Change in Apolipoprotein AI (Apo AI)
Description: Percent change in Apolipoprotein AI (Apo AI) from Baseline (Week 0 of Study 733-005/UP1002) to Week 246 (Week 168 in Study AEGR-733-012).
Time Frame: Baseline and Week 246
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 14
Percent Change | -16.8 (26.62)

53. Secondary Outcome: Percent Change in Apolipoprotein AI (Apo AI)
Description: Percent change in Apolipoprotein AI (Apo AI) from Baseline (Week 0 of Study 733-005/UP1002) to Week 270 (Week 192 in Study AEGR-733-012).
Time Frame: Baseline and Week 270
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent Change | -17.8 (20.12)

54. Secondary Outcome: Percent Change in Apolipoprotein AI (Apo AI)
Description: Percent change in Apolipoprotein AI (Apo AI) from Baseline (Week 0 of Study 733-005/UP1002) to Week 294 (Week 216 in Study AEGR-733-012).
Time Frame: Baseline and Week 294
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide
Number analyzed (Participants) | 3
Percent Change | -30.5 (22.2)

ADVERSE EVENTS:
Time Frame: Week 78 of Study 733-005/UP1002 to Week 294 of Study 733-005/UP1002 (Week 216 of Study AEGR-733-012)
Groups:
- Lomitapide: Maximum tolerated dose of lomitapide (up to 80mg/day) in addition to existing lipid lowering therapy including plasmapheresis or lipid apheresis.
  lomitapide: 5-60 mg po every day
Arm/Group | Lomitapide
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 7/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lomitapide (N=19)
Angina Pectoris (Cardiac disorders) | 1
Aortic Value Incompetence (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Reflux Oesophagitis (Gastrointestinal disorders) | 1
Sudden Cardiac Death (General disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
International Normalized Ratio Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Rhabdomyolsis (Musculoskeletal and connective tissue disorders) | 1
Facial Palsy (Nervous system disorders) | 1
Anticoagulant Therapy (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Arteriovenous Fistula (Vascular disorders) | 1
Hypovolaemic Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lomitapide (N=19)
Anaemia (Blood and lymphatic system disorders) | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 4
Aortic Valve Incompetence (Cardiac disorders) | 1
Chest Pain (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blepharitis (Eye disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 3
Chapped Lips (Gastrointestinal disorders) | 1
Dental Caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 2
Epigastric Discomfort (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Intestinal Mass (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Reflux Oesophagitis (Gastrointestinal disorders) | 1
Stomach Discomfort (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Fatigue (General disorders) | 1
Influenza (General disorders) | 1
Oedema Peripheral (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Vestibulitis (General disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 2
Drug Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Gastrointestinal Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Lower Respiratory Tract Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Sinusitus (Infections and infestations) | 3
Tooth Abscess (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Viral Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint Injury (Injury, poisoning and procedural complications) | 1
Post Procedural Diarrhoea (Injury, poisoning and procedural complications) | 1
Procedural Headache (Injury, poisoning and procedural complications) | 1
Skeletal Injury (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 3
Asparate Aminotransferase Increased (Investigations) | 2
Blood creatine phosphokinase Increased (Investigations) | 1
Blood Potassium Increased (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Carotene Decreased (Investigations) | 1
Carotid Bruit (Investigations) | 1
International Normalized Ratio Decreased (Investigations) | 1
International Normalized Ratio Increased (Investigations) | 1
Liver Function Test Abnormal (Investigations) | 1
Prothrombin Time Prolonged (Investigations) | 1
Transaminases Increased (Investigations) | 1
Vitamin K Decreased (Investigations) | 1
Weight Decreased (Investigations) | 2
White Blood Cell Count Decreased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Iron Deficiency (Metabolism and nutrition disorders) | 1
Oral Intake Reduced (Metabolism and nutrition disorders) | 1
Vitamin E Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Facial Palsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Sensory Disturbance (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Stress (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 1
Anticoagulant Therapy (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Arterial Stenosis (Vascular disorders) | 1
Arteriovenous Fistula (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypovolaemic Shock (Vascular disorders) | 1
Sudden Cardiac Death (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The CTAs generally envision a multisite publication, with the PI's right to publish individually if the pooled publication does not occur within 12 months of study completion. Sponsor has a 45 to 60 day review/approval period to request deletion of confidential information or to request limited deferral to protect its proprietary technology. In one case, the publication provision is more general, specifying that the Sponsor and clinical site will agree on the manner/terms of publication.